CLINICAL TRIAL: NCT05968599
Title: A Real-World Comparison of Clinical Outcomes in Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer (mCRPC) Patients Who Initiated Enzalutamide vs. Abiraterone Acetate (Abiraterone) in Flatiron Electronic Health Record (EHR) Database
Brief Title: A Study to Learn About the Study Medicines Called Enzalutamide and Abiraterone in People With Metastatic Castration-resistant Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: C3431047; NCT05968599 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: metastatic castration-resistant prostate cancer; mCRPC; enzalutamide; abiraterone; overall survival; OS; treatment duration
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — enzalutamide; Abiraterone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Enzalutamide cohort: Patients with mCRPC initiating enzalutamide
  Interventions: Drug: Enzalutamide
- Abiraterone cohort: Patients with mCRPC initiating abiraterone acetate
  Interventions: Drug: Abiraterone acetate

INTERVENTIONS:
Drug: Enzalutamide — As provided in real-world setting
  Other Names: Xtandi
  Groups: Enzalutamide cohort
Drug: Abiraterone acetate — As provided in real-world setting
  Other Names: Yonsa, Zytiga
  Groups: Abiraterone cohort

SUMMARY:
The purpose of this real-world study is to learn about the effects of 2 study medicines called enzalutamide and abiraterone used to treat metastatic castration-resistant prostate cancer (mCRPC).

Prostate cancer is one of the most common cancers in men. The prostate is a gland in the male body that helps make semen. Most prostate cancers need male sex hormones, such as testosterone, to grow. Prostate cancer that keeps growing even when the amount of testosterone in the body is reduced to very low levels is known as "castration-resistant". Metastatic cancer is a cancer that has spread to other parts of the body.

This is a real-world study, not a clinical trial. This means that researchers will look at what happens when men receive the treatments prescribed by their own doctor as part of their usual healthcare treatment. In this study, researchers will use information from the Flatiron Electronic Health Record (EHR) database.

The study will include patients' information from the database for men who:

* Were confirmed by medical tests to have mCRPC
* Started first-line treatment with enzalutamide or abiraterone (index date) for mCRPC
* Had not received chemotherapy treatment before index date
* Were 18 years of age or older on index date

Men who are part of this study will receive enzalutamide or abiraterone as part of their usual treatment for mCRPC.

We will compare the following between men receiving enzalutamide and men receiving abiraterone:

* time from treatment start until death,
* treatment duration, and
* time to next treatment. This study will use patient information from the database until the end of information that is available.

ELIGIBILITY:
Inclusion Criteria:

* Male with metastatic prostate cancer diagnosis and abstracted castration-resistant prostate cancer diagnosis
* Initiated enzalutamide or abiraterone within 14 days prior to or after the metastatic castration-resistant prostate cancer diagnosis. The initiation date of enzalutamide or abiraterone will be defined as the index date.
* At least 18 years old at the index date

Exclusion Criteria:

* Received chemotherapy, novel hormonal therapy, radium-223, olaparib/rucaparib, or immunotherapy prior to the index date
* Had a prior history of other cancers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Men with chemotherapy-naïve mCRPC (aged ≥18 years) who initiated enzalutamide or abiraterone and met eligibility criteria will be included in the study. Patients will be identified from the Flatiron EHR database.
Sampling Method: Non-Probability Sample
Enrollment: 2731 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Up to approximately 8 years
  Overall survival (OS) will be defined as the time from the initiation of enzalutamide or abiraterone to the date of death.

SECONDARY OUTCOMES:
Overall survival among patients without subsequent therapy | Up to approximately 8 years
  Overall survival (OS) among the subgroup of patients who received only enzalutamide without any subsequent therapy or received only abiraterone without any subsequent therapy.
  OS will be defined as the time from the initiation of enzalutamide or abiraterone (i.e., index date) to the date of death.
Treatment duration | Up to approximately 8 years
  Treatment duration will be defined as the time from the initiation of enzalutamide or abiraterone to the discontinuation date. Discontinuation will be defined as the earliest of 1) death, 2) last abstracted end date for enzalutamide or abiraterone, or 3) day before the start of next line of therapy.
Time to subsequent therapy | Up to approximately 8 years
  Time to subsequent therapy will be defined as the time from the initiation of enzalutamide or abiraterone to the start of next line of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3431047